CLINICAL TRIAL: NCT00833898
Title: Psychoeducation For BMT Caregivers: Biobehavioral Markers and Outcome
Brief Title: Stress Management Intervention for Caregivers of Patients Undergoing Bone Marrow Transplant (BMT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-0303; 1R01CA126971-01A1 (NIH)
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Results first posted 2015-09-10 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-11

CONDITIONS: Hematopoietic/Lymphoid Cancer
Keywords: depression; stress; caregiving; anxiety; psychoeducation intervention; psycho-oncology
MeSH Terms: conditions — Hematologic Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caregiver Control (No Intervention): Orientation class; laboratory biomarker analysis; questionnaire administration; survey administration; treatment as usual psychosocial care.
- Caregiver Intervention (Experimental): Orientation class; laboratory biomarker analysis; questionnaire administration; survey administration; Psychoeducation Paced Respiration and Relaxation (PEPRR), which included one-on-one psychoeducation, stress management intervention, with paced respiration.
  Interventions: Device: Paced respiration as part of PEPRR; Behavioral: PEPRR

INTERVENTIONS:
Device: Paced respiration as part of PEPRR — The FDA approved RESPeRATE™ is the size of a portable compact disk (CD) player with a visual display, an elastic belt-type respiratory sensor, and a set of headphones. During a relaxation session, the device analyzes respiratory pattern of the subject and creates a melody of pleasant tones selected by the subject (one for inhalation and one for exhalation). The subjects can observe a cartoon figure on the screen of the device that indicates their inhalation and exhalation. The subject synchronizes their breathing to these tones as the exhalation tone is gradually increased in duration with a target of less than 10 breaths/minute. Subjects were encouraged to use RESPeRATE 3-5 times a week for 20 minutes.
  Other Names: RESPeRATE™
  Arms: Caregiver Intervention
Behavioral: PEPRR — PEPRR consist of 8 sessions, each lasting approximately 60min. The first 4 sessions are weekly, followed by biweekly mtgs for the remaining 4 sessions. Sessions begin the week that the patient receives the transfusion of donor cells. Session 1-4 are conducted at the hospital where the patients receive their transplant. Once discharged from the hospital, sessions will be conducted at the outpatient BMT clinic to coincide with patients' post-transplant visits. Sessions are devoted to a separate topic with the goal of assisting the caregiver in development & application of various stress-mgmt techniques such as effective problem-solving, identifying & challenging cognitive distortions, relaxation techniques, coping skills training, effective use of social support & goal setting.
  Other Names: Psychoeducation & Paced Respiration/Relaxation
  Arms: Caregiver Intervention

SUMMARY:
RATIONALE: A stress management intervention may be more effective than usual care in improving quality of life in caregivers of patients undergoing bone marrow transplant.

PURPOSE: This randomized phase III trial is studying a stress management intervention for caregivers of patients undergoing bone marrow transplant.

DETAILED DESCRIPTION:
Specific Aims

* Further validate a unique saliva collection device in a randomized controlled study of a psychoeducation, paced respiration, and relaxation (PEPRR) intervention for caregivers of patients undergoing bone marrow transplantation.
* Evaluate the suitability of paced respiratory training using RESPeRATE™ for these caregivers.
* Determine the efficacy of a PEPRR intervention on behavioral (stress level, mood and overall health) and physiological (neuroendocrine function, immune function, and sleep) outcomes of these caregivers.

OUTLINE: Caregivers are randomized to 1 of 2 groups.

* Group I (treatment as usual [TAU]): Caregivers and patients attend a 2-hour orientation class that provides an overview of the transplant process, information regarding financial issues and resources that may be available to the patient and caregiver, a review of caregiver duties, dietary restrictions post-transplantation, a brief introduction to stress and stress management, and hands-on training of how to care for a central venous catheter. Patients also receive information in the form of a written manual that provides in-depth information about transplant, including how the transplant works, what to expect, caregiver duties, graft-vs-host disease, and when to contact medical staff for assistance. A voluntary 1-hour weekly caregiver support group is offered on the inpatient BMT unit.
* Group II (psychoeducation, paced respiration, and relaxation [PEPRR]): Caregivers and patients attend a 2-hour orientation class identical to group I. Caregivers also participate in the PEPRR intervention comprising an individualized stress management component and educational component that addresses the psychosocial needs of the caregivers. It also provides self-care and adaptive coping skills. The stress management component addresses caregivers' perception of potential stressors (primary appraisal); perceived ability to control or manage the stressor (secondary appraisal); ability to exert control and cope with the stressor (coping effort); and ongoing evaluation of the stressor and their perceived ability of managing the stressor (reappraisal) and applies coping strategies such as relaxation, prioritizing, goal setting, pacing, and communicating needs. The PEPRR intervention consists of 8 sessions (4 weekly 60-minute sessions followed by 4 biweekly 60-minute sessions) that cover the 100-day period of caregiving post-transplantation. Caregivers also undergo paced respiratory (RESPeRATE™) training for 15 minutes once daily over 12 weeks that measures caregiver adherence and compliance to the relaxation program.

Caregivers and patients undergo psychosocial assessments at approximately 1-3 months prior to randomization and transplantation and again at 1, 3, 6, and 12 months after transplantation. Caregivers also complete questionnaires to assess their stress (PSS, CRA, and IES), mood (POMS, CES-D, and STAI), sleep (PSQI), and health (SF-36).

Caregivers undergo blood and saliva sample collection at baseline and periodically during study for biomarker analysis (e.g., neuroendocrine and immune markers). Caregivers wear an activity watch (actimeter) during each saliva sample collection period.

ELIGIBILITY:
Inclusion Criteria:

* DISEASE CHARACTERISTICS (Meets all of the following criteria):

  * Patient undergoing allogeneic bone marrow transplantation (BMt)
  * Primary caregiver of a BMT patient
  * Has provided care for the patient for at least 50 days of the required 100 days of caregiving following transplant (e.g., 50% of the total time)
* PATIENT CHARACTERISTICS:

  * Able to read and speak English
  * Has telephone access
  * No serious medical condition likely to influence immune and neuroendocrine parameters (caregiver)
  * Alcohol consumption limited to < 2 drinks/day (caregiver)
  * No history of a psychiatric illness unrelated to the experience as a caregiver within the past 18 months (caregiver)
  * No history of a psychiatric illness unrelated to the BMT within the past 18 months (patient)

Exclusion Criteria:

- PRIOR CONCURRENT THERAPY:

• No concurrent steroid medications (caregiver)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2008-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Laudenslager, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Presbyterian/St. Luke's Medical Center (PSLMC) - Denver Midtown, Denver, Colorado

REFERENCES:
- [Background] Simoneau TL, Mikulich-Gilbertson SK, Natvig C, Kilbourn K, Spradley J, Grzywa-Cobb R, Philips S, McSweeney P, Laudenslager ML. Elevated peri-transplant distress in caregivers of allogeneic blood or marrow transplant patients. Psychooncology. 2013 Sep;22(9):2064-70. doi: 10.1002/pon.3259. Epub 2013 Feb 25. PMID 23440998
- [Result] Laudenslager ML, Simoneau TL, Kilbourn K, Natvig C, Philips S, Spradley J, Benitez P, McSweeney P, Mikulich-Gilbertson SK. A randomized control trial of a psychosocial intervention for caregivers of allogeneic hematopoietic stem cell transplant patients: effects on distress. Bone Marrow Transplant. 2015 Aug;50(8):1110-8. doi: 10.1038/bmt.2015.104. Epub 2015 May 11. PMID 25961767
- [Result] Ouseph R, Croy C, Natvig C, Simoneau T, Laudenslager ML. Decreased mental health care utilization following a psychosocial intervention in caregivers of hematopoietic stem cell transplant patients. Ment Illn. 2014 Mar 25;6(1):5120. doi: 10.4081/mi.2014.5120. eCollection 2014 Mar 4. PMID 25478136

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Caregivers and their patients were recruited consecutively between 11/2008 and 4/2012 during pre-transplant screening of all Allo-HSCT patients and their caregivers at a single site (Presbyterian St. Luke's Medical Center, Denver, CO).
Pre-assignment Details: 149 patient-caregiver dyads were consented (298 participants) and 148 dyads were randomized. 1 dyad (2 participants) did not meet the inclusion criteria.
Groups:
- Caregiver Intervention: Orientation class; laboratory biomarker analysis; questionnaire administration; survey administration; Psychoeducation Paced Respiration and Relaxation (PEPRR), includes one-on-one psychoeducation, stress management intervention, with paced respiration.
Period: Overall Study
Arm/Group | Caregiver Control | Caregiver Intervention
Started | 74 | 74
Month 1 (Post Transplantation) | 72 | 74
Month 3 (Post Transplantation) | 66 | 64
Month 6 (Post Transplantation) | 59 | 54
Month 12 (Post Transplantation) | 50 | 50
Completed | 34 | 38
Not Completed | 40 | 36
Not completed — Withdrawal by Subject | 33 | 27
Not completed — Lost to Follow-up | 7 | 7
Not completed — Patient did not receive transplant | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caregiver Control | Caregiver Intervention | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (12.355) | 52.2 (12.169) | 53.5 (12.285)
Gender [Number; unit: participants] — For Caregiver Control gender information, participant did not reported their gender (n = 1).
  participants
    Female | 56 | 56 | 112
    Male | 17 | 18 | 35
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (not Latino/Hispanic) | 68 | 65 | 133
  Black/African-American (not Latino/Hispanic) | 2 | 0 | 2
  Asian/Oriental/Pacific Islander | 0 | 1 | 1
  Latino/Hispanic/Mexian-American | 1 | 6 | 7
  Other | 1 | 1 | 2
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 74 | 74 | 148
Annual income [Number; unit: participants] — Income in dollars
  participants
    < 25,000 | 13 | 11 | 24
    25,000-44,999 | 15 | 14 | 29
    45,000-64,999 | 11 | 15 | 26
    > 65,000 | 31 | 29 | 60
    Unknown or Not Reported | 4 | 5 | 9
Relationship to patient [Number; unit: participants]
  Spouse/partner | 46 | 57 | 103
  Parent | 19 | 8 | 27
  Other | 8 | 8 | 16
  Unknown or Not Reported | 1 | 1 | 2
Employment Status (Before Caregiving) [Number; unit: participants]
  Full-time | 35 | 36 | 71
  Part-time | 11 | 13 | 24
  Unemployed | 8 | 7 | 15
  On leave | 1 | 2 | 3
  Retired | 16 | 13 | 29
  Unknown or Not Reported | 3 | 3 | 6
Employment Status (During Caregiving) [Number; unit: participants]
  Full-time | 16 | 19 | 35
  Part-time | 7 | 10 | 17
  Unemployed | 14 | 8 | 22
  On leave | 17 | 19 | 36
  Retired | 15 | 15 | 30
  Unknown or Not Reported | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Behavioral - Stress Level as Measured by the Perceived Stress Scale (PSS)
Description: The Perceived Stress Scale (PSS) measures the overall level of stress. This instrument contains 14 items accessing overall appraisals of stress in the past month. Minimum score (best value)=0. Maximum score (worst value)=56. A higher score indicates greater stress.
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 4). Caregiver Intervention group: missing responses (n = 2).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 70 | 72
units on a scale
  Baseline | 23.5 [21.6 to 25.3] | 22.7 [20.9 to 24.6]
  Month 1 | 21.6 [19.7 to 23.5] | 22.0 [20.1 to 23.8]
  Month 3 | 23.0 [21.0 to 25.0] | 20.0 [17.9 to 22.0]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.020, Mixed Models Analysis

2. Primary Outcome: Physiological - Cortisol Awakening Response (CAR)
Description: Saliva will be collected using SPIT booklets containing four separate filter papers corresponding to collection times separated by waxed paper. Subjects will be asked to moisten a filter paper 1) immediately after waking, 2) 30 min later, 3) before lunch and 4) 10 hours after waking. They will be asked to collect these samples on three days typical for their schedules at each phase of the. They will indicate the time of each collection. Filters will dry in the booklet. Saliva samples will be aggregated across the three sampling days at each study phase to better reflect the typical pattern for each subject (see Smyth et al, 1997). The change from awakening to 30 minutes in cortisol (CAR) will be characterized by the change between waking and 30 min.
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 15). Caregiver Intervention group: missing responses (n = 15).
Measure: Mean (95% Confidence Interval); unit: ln(nmol/L)
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 59 | 59
ln(nmol/L)
  Baseline | 0.35 [0.23 to 0.48] | 0.25 [0.12 to 0.37]
  Month 1 | 0.33 [0.18 to 0.48] | 0.36 [0.20 to 0.52]
  Month 3 | 0.33 [0.15 to 0.51] | 0.52 [0.34 to 0.70]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.15, Mixed Models Analysis

3. Secondary Outcome: Depression Measured by the Center for Epidemiological Studies Depression Scale (CESD)
Description: The Center for Epidemiological Studies Depression Scale (CES-D) is a self-report 20-item scale designed to measure current depressive symptoms. Scores range from 0-60, with a score at or above 16 reflecting significant depressive symptomatology.
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 5). Caregiver Intervention group: missing responses (n = 2).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 69 | 72
units on a scale
  Baseline | 15.9 [13.7 to 18.1] | 14.6 [12.5 to 16.8]
  Month 1 | 13.8 [11.8 to 15.8] | 13.6 [11.6 to 15.5]
  Month 3 | 16.3 [14.0 to 18.6] | 12.1 [9.8 to 14.5]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.029, Mixed Models Analysis

4. Secondary Outcome: State Anxiety as Measured by the Spielberger State-Trait Anxiety Inventory (STAI)
Description: The State and Trait Anxiety Inventory (STAI) is a validated self-reporting instrument used to assess anxiety in adults. The inventory consists of 2 scales, state anxiety, which evaluates how the subject feels currently (transient anxiety), and trait anxiety, which evaluates how the subject feels generally (general tendency towards anxiety). Each scale consists of 20 questions, and a higher score indicates greater anxiety. Scores range from 20 (no anxiety) to 80 (maximum anxiety).
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 3). Caregiver Intervention group: missing responses (n = 1).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 71 | 73
units on a scale
  Baseline | 42.4 [40.0 to 44.8] | 38.9 [36.6 to 41.3]
  Month 1 | 38.8 [36.4 to 41.2] | 38.0 [35.7 to 40.4]
  Month 3 | 41.6 [38.8 to 44.4] | 34.7 [31.9 to 37.5]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis

5. Secondary Outcome: Total Mood Disturbance (TMD) Score Using the Profile of Mood States (POMS)
Description: POMS stands for the Profile of Mood States. The POMS consists of 65 adjectives rated by subjects on a 5-point scale and six factors that derive from this scale are: 1) tension-anxiety, 2) depression-dejection, 3) anger-hostility, 4) fatigue-inertia, 5) vigor-activity and 6) Confusion-bewilderment. A Total Mood Disturbance (TMD) can be calculated by adding the scores for Tension, Depression, Anger, Fatigue and Confusion and then subtracting the score for Vigour. The range for the Total Mood Disturbance (TMD) score is 0 - 200, with higher score indicating more mood disturbance.
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 4). Caregiver Intervention group: missing responses (n = 1).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 70 | 73
units on a scale
  Baseline | 66.8 [58.9 to 74.8] | 61.0 [53.2 to 68.9]
  Month 1 | 58.0 [50.2 to 65.7] | 59.4 [51.8 to 67.0]
  Month 3 | 65.2 [57.1 to 73.3] | 53.0 [44.8 to 61.2]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis

6. Secondary Outcome: Stress as Measured by Caregiver Burden Using the Caregiver Reaction Assessment (CRA)
Description: The Caregiver Reaction Assessment (CRA) is a measure of caregiver burden. This instrument contains 24 items reflecting the total caregiver situation in the past month. The scale refers to the caregiver. Minimum score (best value)=5. Maximum score (worst value)=25. Higher values reflect the experience of a higher burden.
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 5). Caregiver Intervention group: missing responses (n = 1).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 69 | 73
units on a scale
  Baseline | 10.4 [9.9 to 10.8] | 10.2 [9.7 to 10.6]
  Month 1 | 10.8 [10.2 to 11.4] | 10.8 [10.3 to 11.4]
  Month 3 | 10.9 [10.3 to 11.5] | 10.6 [9.9 to 11.2]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.40, Mixed Models Analysis

7. Secondary Outcome: Sleep as Assessed by the Pittsburgh Sleep Quality Inventory (PSQI) Total Score
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-rated scale to measure quality of sleep via questions regarding sleep latency, duration, efficiency, disturbances, use of sleep medication, and daytime dysfunction. Scores range from 0 to 21, where scores greater than 5 indicate poor sleep quality.
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 3). Caregiver Intervention group: missing responses (n = 1).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 71 | 73
units on a scale
  Baseline | 11.1 [10.4 to 11.7] | 11.4 [10.8 to 12.1]
  Month 1 | 11.2 [10.6 to 11.9] | 11.2 [10.6 to 11.9]
  Month 3 | 11.2 [10.5 to 11.9] | 11.0 [10.3 to 11.7]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.44, Mixed Models Analysis

8. Secondary Outcome: Mental Component Summary Via the Short-Form 36-Item Health Survey Version 2.0 (SF-36M)
Description: The Short-Form 36-Item Health Survey Version 2.0 (SF-36) is 36-item form related to 8 health concepts (physical functioning, role physical, role emotional, general health, social functioning, bodily pain, vitality, mental health) and 2 summary scores (physical and mental component summary). Role emotional, social functioning and mental health contribute to mental component; as well as the social functioning, vitality, and general health. Scores are based on a scale from 0 to 100, with higher scores defining more favorable health state.
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 4). Caregiver Intervention group: missing responses (n = 4).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline | 42.7 [40.1 to 45.3] | 45.1 [42.6 to 47.7]
  Month 1 | 43.8 [41.0 to 46.6] | 45.7 [42.9 to 48.4]
  Month 3 | 43.5 [40.6 to 46.4] | 47.0 [43.9 to 50.0]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.75, Mixed Models Analysis

9. Secondary Outcome: Physical Component Summary Via the Short-Form 36-Item Health Survey Version 2.0 (SF-36P)
Description: The Short-Form 36-Item Health Survey Version 2.0 (SF-36) is 36-item form related to 8 health concepts (physical functioning, role physical, role emotional, general health, social functioning, bodily pain, vitality, mental health) and 2 summary scores (physical and mental component summary). Physical functioning, role physical and bodily pain contribute to physical component; as well as the social functioning, vitality, and general health. Scores are based on a scale from 0 to 100, with higher scores defining more favorable health state.
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 4). Caregiver Intervention group: missing responses (n = 4).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline | 53.8 [51.9 to 55.7] | 54.7 [52.8 to 56.6]
  Month 1 | 54.0 [51.7 to 56.3] | 52.9 [50.6 to 55.2]
  Month 3 | 53.7 [51.6 to 55.8] | 54.0 [51.8 to 56.1]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.17, Mixed Models Analysis

10. Secondary Outcome: Stress as Measured by the Impact of Events Scale (IES)
Description: The Impact of Events Scale (IES), a widely accepted measure for evaluating intrusive thoughts regarding an event or situation. The scale consists of 15 items (7 measuring intrusive thoughts and 8 measuring avoidance) scored on a 5-point Likert Scale. Minimum score (best value)=0. Maximum score (worst value)=75. Scores over 20 indicate significant levels of PTS-like symptoms. The IES is anchored to the caregiving experience.
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 4). Caregiver Intervention group: missing responses (n = 2).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 70 | 72
units on a scale
  Baseline | 31.4 [29.5 to 33.3] | 29.8 [27.9 to 31.7]
  Month 1 | 31.0 [29.0 to 33.0] | 29.1 [27.1 to 31.1]
  Month 3 | 30.3 [28.0 to 32.6] | 28.4 [26.1 to 30.8]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.97, Mixed Models Analysis

11. Secondary Outcome: The Slope of the Diurnal Decline in Salivary Cortisol (SlopeC)
Description: The SlopeC has been noted to be affected by stressful experiences. From diurnal saliva collections at each phase we will fit curves between awake, before lunch, and 10 hours after awaking to characterize the diurnal change in salivary cortisol (SlopeC).
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 12). Caregiver Intervention group: missing responses (n = 12).
Measure: Mean (95% Confidence Interval); unit: ln[(nmol/L)/hour]
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 62 | 62
ln[(nmol/L)/hour]
  Baseline | -0.12 [-0.15 to -0.08] | -0.12 [-0.16 to -0.09]
  Month 1 | -0.10 [-0.13 to -0.07] | -0.12 [-0.15 to -0.08]
  Month 3 | -0.12 [-0.15 to -0.10] | -0.11 [-0.14 to -0.09]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.55, Mixed Models Analysis

12. Secondary Outcome: The Slope of the Diurnal Decline (SlopeD) in Salivary Dehydroepiandrosterone (DHEA)
Description: The SlopeD has been noted to be affected by affective disorders such as depression. From diurnal saliva collections at each phase we will fit curves between awake, before lunch, and +10 hours after awaking to characterize the diurnal change in salivary DHEA.
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 16). Caregiver Intervention group: missing responses (n = 15).
Measure: Mean (95% Confidence Interval); unit: ln[(nmol/L)/hour]
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 58 | 59
ln[(nmol/L)/hour]
  Baseline | -0.11 [-0.14 to -0.09] | -0.13 [-0.15 to -0.10]
  Month 1 | -0.13 [-0.16 to -0.10] | -0.15 [-0.18 to -0.12]
  Month 3 | -0.13 [-0.15 to -0.11] | -0.17 [-0.18 to -0.15]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.30, Mixed Models Analysis

13. Secondary Outcome: Area Under the Curve for Salivary Cortisol (AUCc)
Description: The AUCc will be determined between awaking, 30 minutes after awaking, prior to lunch, and 10 hours after awaking from saliva samples collected using a special filter collection device applied in this study. This area will be an estimate of total cortisol released during this time period.
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 16). Caregiver Intervention group: missing responses (n = 14).
Measure: Mean (95% Confidence Interval); unit: ln[(nmol/L)*hour]
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 58 | 60
ln[(nmol/L)*hour]
  Baseline | 3.85 [3.71 to 3.99] | 3.65 [3.51 to 3.79]
  Month 1 | 3.78 [3.61 to 3.96] | 3.80 [3.62 to 3.98]
  Month 3 | 3.77 [3.55 to 3.99] | 3.68 [3.45 to 3.91]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.67, Mixed Models Analysis

14. Secondary Outcome: Area Under the Curve for Salivary DHEA (AUCd)
Description: The AUCd will be determined between awaking, 30 minutes after awaking, prior to lunch, and 10 hours after awaking from saliva samples collected using a special filter collection device applied in this study. This area will be an estimate of total DHEA released during this time period.
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 16). Caregiver Intervention group: missing responses (n = 14).
Measure: Mean (95% Confidence Interval); unit: ln[(nmol/L)*hour]
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 58 | 60
ln[(nmol/L)*hour]
  Baseline | 1.44 [1.26 to 1.62] | 1.64 [1.46 to 1.81]
  Month 1 | 1.52 [1.34 to 1.70] | 1.41 [1.23 to 1.59]
  Month 3 | 1.56 [1.37 to 1.74] | 1.35 [1.16 to 1.54]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis

15. Secondary Outcome: Host Defense Assessed by Natural Killer (NK) Cell Cytotoxicity
Description: The activity of natural killer (NK) cells is modified by psychosocial and behavioral states (Cacioppo et al., 1998; Irwin et al., 1991; Kiecolt-Glaser et al., 1991; Kiecolt-Glaser, 1999; Kiecolt-Glaser, McGuire, Robles, et al., 2002a; Kiecolt-Glaser, McGuire, Robles, et al., 2002b). Natural cytotoxicity will be determined toward K562 target cell lines as previously described (Laudenslager et al., 1998; Scanlan, et al., 1995). Percent lysis at each effector to target ratio will be found from the median value of each triplicate determination and from which the percent lysis/NK + cell will be determined for 20% lysis (lytic units/NK+ cell).
Time Frame: Baseline (prior to transplant), 1 and 3 post transplant
Population: Caregiver Control group missing responses (n = 8). Caregiver Intervention group: missing responses (n = 2).
Measure: Mean (95% Confidence Interval); unit: ln(% Lysis/NK+ Cell)
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 66 | 72
ln(% Lysis/NK+ Cell)
  Baseline | -1.01 [-1.23 to -0.78] | -1.07 [-1.29 to -0.86]
  Month 1 | -1.09 [-1.28 to -0.89] | -1.17 [-1.37 to -0.97]
  Month 3 | -1.09 [-1.32 to -0.86] | -1.27 [-1.49 to -1.04]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.80, Mixed Models Analysis

16. Secondary Outcome: Plasma C-reactive Protein (CRP)
Description: Plasma c-reactive (CRP) is an acute phase reactant that has been found to be predictive of cardiovascular disease. Is is also an inflammatory marker that will be assessed using high sensitivity CRP assays.
Time Frame: Baseline (prior to transplant) and 3 post transplant
Population: Caregiver Control group missing responses (n = 7). Caregiver Intervention group: missing responses (n = 6).
Measure: Mean (95% Confidence Interval); unit: ln(mg/L)
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 67 | 68
ln(mg/L)
  Baseline | 0.18 [-0.16 to 0.51] | 0.27 [-0.06 to 0.61]
  Month 3 | 0.03 [-0.37 to 0.43] | -0.10 [-0.50 to 0.30]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.26, Mixed Models Analysis

17. Secondary Outcome: Plasma Inflammatory Marker Interleukin 1 Beta (IL-1 Beta)
Description: Inflammatory markers increase in association with stress. IL-1 beta is an inflammatory marker that will be determined in plasma using multiplex array technology.
Time Frame: Baseline (prior to transplant) and 3 post transplant
Population: Wilcoxon signed rank t-test
Measure: Median (Standard Deviation); unit: pg/mL
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 43 | 45
pg/mL
  Baseline | .39 (.62) | .39 (.73)
  3 Months | .39 (.70) | .39 (.22)
Statistical Analysis 1: Comparison: Caregiver Control; Test type: Superiority or Other; p = .58, Wilcoxon (Mann-Whitney) — P-values represent separate wilcoxon paired sample signed rank test
Statistical Analysis 2: Comparison: Caregiver Intervention; Test type: Superiority or Other; p = .33, Wilcoxon (Mann-Whitney) — P-values represent separate wilcoxon paired sample signed rank test

18. Secondary Outcome: Plasma Inflammatory Marker Interleukin 6 (IL-6)
Description: Inflammatory markers increase in association with stress. IL-6 is an inflammatory marker that will be assessed using high sensitivity IL-6 assays.
Time Frame: Baseline (prior to transplant) and 3 post transplant
Population: Caregiver Control group missing responses (n = 11). Caregiver Intervention group: missing responses (n = 4).
Measure: Mean (95% Confidence Interval); unit: ln(pg/mL)
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 63 | 70
ln(pg/mL)
  Baseline | -0.33 [-0.54 to -0.13] | -0.56 [-0.76 to -0.37]
  Month 3 | -0.13 [-0.34 to 0.07] | -0.45 [-0.65 to -0.25]
Statistical Analysis 1: Comparison: Caregiver Control vs Caregiver Intervention; Test type: Superiority or Other; p = 0.53, Mixed Models Analysis

19. Secondary Outcome: Plasma Inflammatory Marker Interleukin 4 (IL-4)
Description: Inflammatory markers increase in association with stress. IL-4 is an anti inflammatory marker that will be determined in plasma using multiplex array technology.
Time Frame: Baseline (prior to transplant) and 3 post transplant
Population: Wilcoxon signed rank t-test
Measure: Median (Standard Deviation); unit: pg/mL
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 43 | 45
pg/mL
  Baseline | 1.56 (1.29) | 1.56 (0.00)
  3 months | 1.56 (4.02) | 1.56 (0.00)
Statistical Analysis 1: Comparison: Caregiver Control; Test type: Superiority or Other; p = .18, Wilcoxon (Mann-Whitney) — P-values represent separate wilcoxon paired sample signed rank test
Statistical Analysis 2: Comparison: Caregiver Intervention; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney) — P-values represent separate wilcoxon paired sample signed rank test

20. Secondary Outcome: Plasma Inflammatory Marker Interleukin 10 (IL-10)
Description: Inflammatory markers increase in association with stress. IL-10 is an anti inflammatory marker that will be determined in plasma using multiplex array technology.
Time Frame: Baseline (prior to transplant) and 3 post transplant
Population: Wilcoxon signed rank t-test
Measure: Median (Standard Deviation); unit: pg/mL
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 43 | 45
pg/mL
  Baseline | 1.72 (3.50) | 1.60 (1.19)
  3 months | 1.60 (2.69) | 1.60 (1.33)
Statistical Analysis 1: Comparison: Caregiver Control; Test type: Superiority or Other; p = .43, Wilcoxon (Mann-Whitney) — P-values represent separate wilcoxon paired sample signed rank test
Statistical Analysis 2: Comparison: Caregiver Intervention; Test type: Superiority or Other; p = .72, Wilcoxon (Mann-Whitney) — P-values represent separate wilcoxon paired sample signed rank test

21. Secondary Outcome: Plasma Inflammatory Marker Tumor Necrosis Factor (TNF)
Description: Inflammatory markers increase in association with stress. TNF is an inflammatory marker that will be determined in plasma using multiplex array technology.
Time Frame: Baseline (prior to transplant) and 3 post transplant
Population: Wilcoxon signed rank t-test
Measure: Median (Standard Deviation); unit: pg/mL
Arm/Group | Caregiver Control | Caregiver Intervention
Number analyzed (Participants) | 43 | 45
pg/mL
  Baseline | 4.70 (5.29) | 4.70 (2.01)
  3 months | 4.70 (5.37) | 4.70 (2.69)
Statistical Analysis 1: Comparison: Caregiver Control; Test type: Superiority or Other; p = .43, Wilcoxon (Mann-Whitney) — P-values represent separate wilcoxon paired sample signed rank test
Statistical Analysis 2: Comparison: Caregiver Intervention; Test type: Superiority or Other; p = .72, Wilcoxon (Mann-Whitney) — P-values represent separate wilcoxon paired sample signed rank test

ADVERSE EVENTS:
Arm/Group | Caregiver Control | Caregiver Intervention
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No